CLINICAL TRIAL: NCT04197115
Title: Difference in Mortality and Evolution in Septic Patients Treated With Vitamin C, Tiamine, Cyanocobalamine, Pyridoxine and Hydrocortisone Treated at the ICU of General Hospital Zone 11 IMSS Piedras Negras Coahuila.
Brief Title: Vitamin C, Thiamine, Cyanocobalamine, Pyridoxine and Hydrocortisone in Sepsis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IMSS Hospital General de Zona 11, Piedras Negras (Other)
Responsible Party: Principal Investigator, JOSE IVAN RODRIGUEZ DE MOLINA SERRANO, Head of Intensive Care Unit Jose Ivan RodriguezdeMolina Critical Care Ph., IMSS Hospital General de Zona 11, Piedras Negras
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: F-2019-506-010
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Sepsis; Septic Shock
Keywords: sepsis; septic shock; Vitamin C; Hydrocortisone; Mortality
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Ascorbic Acid; Hydrocortisone; Hydroquinones; Vitamin B Complex

STUDY DESIGN:
Intervention Model Description: Prospective longitunal experimental
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 (No Intervention): Septic patients admited to ICU whick will be treated as specified in current guidelines.
- Phase 2 (Active Comparator): Septic patients admitted to ICU which will be treated as specified in current guidelines adding:
  Vitamin C Hydrocortisone B complex (Thiamine 100mg, Pyridoxine 5 mg and Cyanocobalamin 50 mcg)
  Interventions: Drug: Vitamin C; Drug: Hydrocortisone; Drug: Complex B

INTERVENTIONS:
Drug: Vitamin C — Intravenous vitamin C (1.5 grams every 6 hours) will be administered for 4 days or until ICU discharge.
  Other Names: ascorbic acid
  Arms: Phase 2
Drug: Hydrocortisone — Intravenous hydrocortisone (50 mg every 6 hours) will be administered for 4 days or until ICU discharge.
  Other Names: Hydrocortisone sodium succinate
  Arms: Phase 2
Drug: Complex B — Complex B ((Thiamine 100mg, Pyridoxine 5 mg and Cyanocobalamin 50 mcg) 1 tablet enteral route every 6 horas for 4 days or until ICU discharge
  Other Names: vitamin B complex
  Arms: Phase 2

SUMMARY:
Prospective, experimental, longitudinal cohort study in septic patients treated at ER and ICU at General Hospital Zone 11 IMSS Piedras Negras Coahuila.

Interventions, will be implementd in 2 consecutive periods of 6 months Phase 1: 6 months period, septic patients treated only with standard treatment.

Phase 2: 6 months period, septic patients treated with Vitamin C, Thiamine, Cyanocobalamine, Pyridoxine and Hydrocortisone + standard treatment.

DETAILED DESCRIPTION:
The research protocol will consist of two phases:

Phase 1: collection of statistical data of septic patients in whom standard treatment will be applied according to clinical practice guidelines, with an approximate duration of 6 months

Phase 2: experimental period lasting 6 months in which the standard treatment will be applied according to clinical practice guidelines + the treatment protocol consisting of Vitamin C 1.5 g IV every 6 hours, Hydrocortisone 50 mg IV every 6 hours and in case of having Enteral route Complex B (Thiamine 100 mg, Pyridoxine 5 mg, Cyanocobalamin 50 mcg) 1 tablet every 6 hours for 4 continuous days or until discharge from the ICU patient.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or confirmed infection as evidenced by ordering of blood cultures and administration of at least one antimicrobial agent
* Acute respiratory or cardiovascular organ dysfunction attributed to sepsis as evidenced by at least one of the following requirements:
* Vasopressor Requirement - Continuous infusion of norepinephrine, epinephrine, vasopressin, dopamine, phenylephrine or other vasopressor agents at any dose for greater than 1 hour and required to maintain a mean arterial pressure ≥ 65 mm Hg despite intravenous crystalloid infusion of at least 1000cc
* Respiratory Support Requirement - Acute hypoxemic respiratory failure defined as persistent hypoxemia ( partial pressure of arterial oxygen (PaO2)/fraction of inspired oxygen (FiO2) ≤ 300 or blood oxygen saturation (SpO2)/FiO2 ≤ 315) requiring (1) intubation and mechanical ventilation, or (2) positive pressure ventilation via tight- fitting f ace mask (i.e. continuous positive airway pressure (CPAP) or bilevel positive airway pressure (BiPAP) or (3) high flow nasal cannula ≥ 45 liter per minute (LPM) flow and FiO2

  * 0.40
* Anticipated or confirmed intensive care unit (ICU) admission

Exclusion Criteria:

* Organ dysfunction present > 24 hours at time of enrollment
* Limitations of care (defined as refusal of cardiovascular and respiratory support modes described in inclusion criteria 7.1.b) including "do not intubate" (DNI) status
* Current hospitalization > 30 days at time of randomization
* Chronic hypoxemia requiring supplemental non-invasive oxygen (nasal cannula or NIPPV) or home mechanical ventilation
* Chronic cardiovascular failure requiring home mechanical hemodynamic support (e.g., LVAD) or home chemical hemodynamic support (e.g., milrinone)
* Known allergy or contraindication to vitamin C, thiamine, and/or corticosteroids (including previously or currently diagnosed primary hyperoxaluria and/or oxalate nephropathy, or nown/suspected ethylene glycol ingestion, or known glucose-6-phosphate dehydrogenase (G6PD) deficiency)
* Currently receiving intravenous vitamin C as a treatment for sepsis OR any dose of vitamin C exceeding 1 gram daily
* Chronic disease/illness that, in the opinion of the site investigator, have an expected lifespan of < 30 days unrelated to current sepsis diagnosis (e.g., stage IV malignancy, neurodegenerative disease, etc.)
* Pregnancy or known active breastfeeding
* Prisoner or Incarceration
* Current participation in another interventional pharmaceutical research study for sepsis Inability or unwillingness of subject or legal surrogate/representative to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Difference in hospital mortality in phase 1 vs phase 2 groups | 1 year
  Quantitative variable: Metric unit: number (percentage); Mortality in hospital
Difference in Intensive Care Unit Mortality in phase 1 vs phase 2 groups | 1 year
  Quantitative variable; Metric unit: number (percentage); Mortality in Intensive Care Unit

SECONDARY OUTCOMES:
Difference in SOFA (Sequential Organ Failure Assessment) between phase 1 vs phase 2 groups | 1 year
  Quantitative variable: Maximal score of SOFA (Sequential Organ Failure Assessment) will be recorded; Value range 0-24 points.
Difference in number of days with vasopressor use between phase 1 vs phase 2 groups. | 1 year
  Quantitative variable; Metric unit: number of days with vasopressors; Vasopressors defined as use of at leas one or in addition of epinephrine, norepinephrine, dobutamine, dopamine, vasopressin.

CONTACTS AND LOCATIONS:
Overall Officials: JOSE IVAN RODRIGUEZ DE MOLINA SERRANO, MD, Principal Investigator — IMSS HGZ 11 UTI PIEDRAS NEGRAS COAHUILA MEXICO
Locations (1):
- Hospital General Zona 11 Imss Piedras Negras Coahuila, Piedras Negras, Coahuila, Mexico

IPD SHARING:
Plan to Share IPD: No